CLINICAL TRIAL: NCT00660543
Title: Early Assessment of Tumor Response to Therapy Using Ferumoxytol (Code 7228) as an MR Contrast Agent in Patients With Glioblastoma Multiforme (MedDRA Code 10018337)
Brief Title: MRI Study With Ferumoxytol in Assessing Early Response in Patients With Glioblastoma Multiforme Receiving Temozolomide and Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Edward Neuwelt, Professor, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00002753; NCI-2015-00224 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SOL-06062-LX; 813; NCI-2015-00204; 8097; 2753 (Other: OHSU Knight Cancer Institute); P30CA069533 (NIH)
Record Dates: First submitted 2008-04-10; First posted 2008-04-17 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Adult Brain Glioblastoma
MeSH Terms: interventions — Gadolinium; Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ferumoxytol (Experimental): Patients receive ferumoxytol non-stoichiometric magnetite IV on day 2 then undergo DSC MRI, and DCE MRI, DWI (day 1 only), and TOF MR angiography on days 1-3 at 4 time points: before radiation, 3 weeks after initiation of radiation plus temozolomide, at the end of radiation (6 weeks post first dose) and 6 weeks after radiation (12 weeks post first dose). Ferumoxytol non-stoichiometric magnetite administration continues in the absence of unacceptable toxicity.
  Interventions: Drug: Ferumoxytol Non-Stoichiometric Magnetite; Other: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Other: Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging; Other: Diffusion Weighted Imaging; Other: MRI-Based Angiogram
- Gadoteridol (Active Comparator): Patients receive gadoteridol IV on day 1 then undergo DSC MRI, and DCE MRI, DWI (day 1 only), and TOF MR angiography on days 1-3 at 4 time points: before radiation, 3 weeks after initiation of radiation plus temozolomide, at the end of radiation (6 weeks post first dose) and 6 weeks after radiation (12 weeks post first dose).
  Interventions: Drug: Gadolinium; Other: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Other: Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging; Other: Diffusion Weighted Imaging; Other: MRI-Based Angiogram
- Gadoteridol Leakage Corrected (Active Comparator): Patients receive gadoteridol IV on day 1 then undergo DSC MRI, and DCE MRI, DWI (day 1 only), and TOF MR angiography on days 1-3 at 4 time points: before radiation, 3 weeks after initiation of radiation plus temozolomide, at the end of radiation (6 weeks post first dose) and 6 weeks after radiation (12 weeks post first dose).
  Interventions: Drug: Gadolinium; Other: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Other: Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging; Other: Diffusion Weighted Imaging; Other: MRI-Based Angiogram

INTERVENTIONS:
Drug: Gadolinium — Given IV
  Other Names: Gd
  Arms: Gadoteridol; Gadoteridol Leakage Corrected
Drug: Ferumoxytol Non-Stoichiometric Magnetite — Given IV
  Other Names: Fe3O4; Feraheme; Ferumoxytol
  Arms: Ferumoxytol
Other: Dynamic Contrast-Enhanced Magnetic Resonance Imaging — Undergo DCE MRI
  Other Names: DCE MRI; DCE-MRI
Other: Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging — Undergo DSC MRI
  Other Names: DSC-MRI; Dynamic Susceptibility Contrast-Enhanced MRI
Other: Diffusion Weighted Imaging — Undergo DWI
  Other Names: Diffusion Weighted MRI; DWI; DWI MRI; DWI-MRI
Other: MRI-Based Angiogram — Undergo TOF MR angiography
  Other Names: Magnetic Resonance Angiogram; MRA

SUMMARY:
This pilot clinical trial studies how a magnetic resonance imaging (MRI) study with ferumoxytol works as a contrasting agent in assessing early response in patients with glioblastoma multiforme receiving temozolomide and radiation therapy. Ferumoxytol is a very small form of iron particles that are injected into the body and taken up by certain tissues which may make these tissues easier to see during imaging. Diagnostic procedures, such as an MRI study with ferumoxytol, may help measure a patient's response to earlier treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize glioblastoma multiforme (GBM) tumor vascular properties using ferumoxytol (ferumoxytol non-stoichiometric magnetite) and compare to those obtained using gadolinium (Gd) based MRI contrast agent.

II. To characterize vascular changes in GBM tumors associated with standard radio/chemotherapy.

SECONDARY OBJECTIVES:

I. Cerebral blood flow (CBF), mean transit time (MTT), and time-to-peak (TTP) perfusion parameters will be measured for each contrast agent and evaluated in post-hoc analysis.

II. To obtain qualitative assessment of tumor vascularity using time-of-flight (TOF) magnetic resonance (MR) angiography techniques.

III. To characterize changes in the apparent diffusion coefficient (ADC) of tumor water associated with standard radio/chemotherapy in GBM.

OUTLINE:

Patients receive gadolinium intravenously (IV) on day 1 and ferumoxytol non-stoichiometric magnetite IV on day 2 then undergo dynamic susceptibility contrast enhanced (DSC) MRI, and dynamic contrast enhanced (DCE) MRI, diffusion-weighted imaging (DWI) (day 1 only), and TOF MR angiography on days 1-3 at 4 time points: before radiation, 3 weeks after initiation of radiation plus temozolomide, at the end of radiation (6 weeks post first dose) and 6 weeks after radiation (12 weeks post first dose). Ferumoxytol non-stoichiometric magnetite administration continues in the absence of unacceptable toxicity. Patients also receive temozolomide and undergo radiation therapy per standard of care.

After completion of ferumoxytol non-stoichiometric magnetite administration, patients are followed up for 4-6 weeks and then periodically until the resolution or stabilization of unacceptable toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have radiologically and histologically confirmed diagnosis of glioblastoma multiforme
* Patients must have measurable disease, defined as evident tumors with gadolinium enhancement on MRI that is measurable in at least one diameter and visible on both axial and sagittal or coronal views
* Life expectancy of greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 50%)
* Patients scheduled for standard therapy (6 weeks radiation therapy (RT) ~ 60 Gy, plus temozolomide 75 mg/m^2 during 6 week [w] RT, and followed routine monthly temozolomide therapy)
* Patients must be on a stable or decreasing dose (up to 8 mg daily) of dexamethasone throughout the study
* After entry into the study, patients are expected to be followed for at least 1 month after the last infusion of ferumoxytol
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document; all patients, or their legal guardians, must sign a written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization in accordance with institutional guidelines

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ferumoxytol: parenteral iron, parenteral dextran, parenteral iron-dextran, or parenteral iron-polysaccharide preparations (Ferumoxytol Investigator's Drug Brochure, 2005); patients with significant drug or other allergies or autoimmune diseases may be enrolled at the Investigator's discretion
* Patients with clinically significant signs of uncal herniation, such as acute pupillary enlargement, rapidly developing motor changes (over hours), or rapidly decreasing level of consciousness, are not eligible
* Patients who require monitored anesthesia for MRI scanning
* Patients with history of hemochromatosis or iron overload
* Patients with renal insufficiency (glomerular filtration rate (GFR) < 50)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with ferumoxytol
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Neuwelt, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Gadoteridol + Ferumoxytol Contrast Agent: Subjects all received gadolinium enhanced MR on day 1, ferumoxytol enhanced MR on day 2, and delayed MR imaging on day 3 - this 3 day sequence of imaging was repeated at four time points.
Period: Overall Study
Arm/Group | Gadoteridol + Ferumoxytol Contrast Agent
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gadoteridol + Ferumoxytol Contrast Agent
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 60 [43 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Mean Cerebral Blood Volume (CBV)
Description: Radiographical progression is determined based on RANO criteria.
Time Frame: At radiographical progression (between 6 and 12 weeks post first dose of chemoradiation)
Population: All patients with treated GMB showed apparent tumor progression on conventional MR images.
Measure: Mean (Standard Deviation); unit: mL/g
Groups:
- Ferumoxytol: Patients receive gadolinium IV on day 1 and ferumoxytol non-stoichiometric magnetite IV on day 2 then undergo DSC MRI, and DCE MRI, DWI (day 1 only), and TOF MR angiography on days 1-3 at 4 time points: before radiation, 3 weeks after initiation of radiation plus temozolomide, at the end of radiation (6 weeks post first dose) and 6 weeks after radiation (12 weeks post first dose).
- Gadoteridol Leakage Correction: Patients receive gadoteridol IV on day 1 then undergo DSC MRI, and DCE MRI, DWI (day 1 only), and TOF MR angiography on days 1-3 at 4 time points: before radiation, 3 weeks after initiation of radiation plus temozolomide, at the end of radiation (6 weeks post first dose) and 6 weeks after radiation (12 weeks post first dose).
Arm/Group | Ferumoxytol | Gadoteridol | Gadoteridol Leakage Correction
Number analyzed (Participants) | 14 | 14 | 14
mL/g | 2.5 (2.1) | 1.38 (1.73) | 2.36 (1.94)
Statistical Analysis 1: Comparison: Ferumoxytol vs Gadoteridol; Test type: Superiority or Other; p = .003, t-test, 1 sided; Differences between groups were assessed by using the Student paired t test and were graphed by using Bland-Altman plots
Statistical Analysis 2: Comparison: Ferumoxytol vs Gadoteridol Leakage Correction; Test type: Superiority or Other; p = .008, t-test, 1 sided; [statistical method as in outcome 1, analysis 1]

2. Primary Outcome: Tumor Progression on Conventional MR
Description: Tumor progression was assessed by RANO criteria (Wen, 2010).
Time Frame: Anytime between baseline and 12 weeks post treatment initiation: average 6 weeks post treatment initiation.
Measure: Number; unit: participants
Groups:
- Tumor Progression on Conventional MR: Tumor progression was assessed by RANO criteria (Wen, 2010).
Arm/Group | Tumor Progression on Conventional MR
Number analyzed (Participants) | 14
participants | 14

ADVERSE EVENTS:
Groups:
- Ferumoxytol: Subjects all received ferumoxytol enhanced MR on day 1, ferumoxytol enhanced MR on day 2, and delayed MR imaging on day 3 - this 3 day sequence of imaging was repeated at four time points
- Gadoteridol; Gadoteridol With Leakage Correction: Subjects all received gadolinium enhanced MR on day 1, ferumoxytol enhanced MR on day 2, and delayed MR imaging on day 3 - this 3 day sequence of imaging was repeated at four time points
Arm/Group | Ferumoxytol | Gadoteridol | Gadoteridol With Leakage Correction
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 0/14 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferumoxytol (N=14) | Gadoteridol (N=14) | Gadoteridol With Leakage Correction (N=14)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No